CLINICAL TRIAL: NCT05882617
Title: Assessment of Patient Satisfaction in Completely Edentulous Patients Receiving Removable Implant Overdentures Retained by Different Numbers of Implants .A Randomized Clinical Trial
Brief Title: Patient Satisfaction With Different Numbers of Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed awaad, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 33922
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: three parallel arms one comparator and two interventions
Who Masked: Outcomes Assessor
Masking Description: only statistician was masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental (Experimental): single impalnts supported overdenture
  Interventions: Other: implants supported overdentures
- active comparator (Active Comparator): two implants supported overdenture
  Interventions: Other: implants supported overdentures
- others (Other): four implants supported overdenture
  Interventions: Other: implants supported overdentures

INTERVENTIONS:
Other: implants supported overdentures — implant supported and retained with different number of implants retained by ball attachments

SUMMARY:
the goal of this randomized controlled trial aimed to assess patient satisfaction for completely edentulous patients with implant overdenture retained by ball attachment over a single symphyseal , or four interforaminal implants when compared to two interforaminal ones

DETAILED DESCRIPTION:
48 edentulous patients were recruited and randomized to receive either 1,2 or 4 implants for a mandibular overdenture,3 months later implants were uncovered, and ball attachments were torqued, and all overdentures were picked up ,patient satisfaction questionnaires were recorded for all patients 2 weeks after pickup 3 months ,6 months, 9 months and 1year.

ELIGIBILITY:
Inclusion criteria

* completely edentulous patients with restorative space of 12-15 mm,
* keratinized gingiva of 5 mm

Exclusion criteria

* Exclusion Criteria:
* uncontrolled diabetes
* bruxers
* smokers

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
patient satisfaction for masticatory ability, mental life comfortability with dentures | one year
  A translated into Arabic form of patient satisfaction questionnaire to match the language and environmental background of the patients was answered by all subjects, Each response was given a score range from 0 to 4 where zero represents the best result . Questionnaire was divided into three categories questions, the first section was a direct questions to the patient answered by one of some choices, and each choice had a number which will be summed up and giving a score, The second section was a visual answered question; in which patient chose from best to worst on a given scale. The marked point will be translated into a number from zero (the best) to ten (the worst). The third section was a YES/ NO questions, answered shortly by the patient in the terms of yes or No.
  A translated into Arabic form of patient satisfaction questionnaire to match the language and environmental background of the patients was answered by all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Elkady phd, Study Director — lecturer
Locations (2):
- Egypt (2):
  - Doaa Mahmoud Elkady, Cairo
  - Nesma Mohamed Awaad, Cairo

IPD SHARING:
Plan to Share IPD: No